CLINICAL TRIAL: NCT05266417
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase II Study to Evaluate the Safety, Tolerability, and Efficacy of Intranasal Insulin and Glutathione as an Add-On Therapy in Subjects With Parkinson's Disease (NOSE-PD)
Brief Title: Intranasal Insulin and Glutathione as an Add-On Therapy in Parkinson's Disease
Acronym: NOSE-PD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gateway Institute for Brain Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-GTY-008-01
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
Keywords: Insulin; Glutathione; Intranasal
MeSH Terms: conditions — Parkinson Disease; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active (Experimental): Insulin (Novolin R) and Glutathione (INS-GSH)
  Interventions: Drug: INS-GSH
- Control (Placebo Comparator): Placebo
  Interventions: Drug: Matched Placebos

INTERVENTIONS:
Drug: INS-GSH — Intranasal INS-GSH Twice Daily
  Arms: Active
Drug: Matched Placebos — Intranasal Matched Placebos Twice Daily
  Other Names: Insulin Matched Placebo and Glutathione Matched Placebo
  Arms: Control

SUMMARY:
This study will be evaluating the safety and efficacy of insulin and glutathione in subjects with Parkinson's Disease compared to placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* Documented clinical diagnosis of idiopathic PD
* Modified HY stage < 5
* Able to administer study drug or have a caregiver throughout the duration of the study to help administer drug
* Willing to continue diet, exercise and medications reported at baseline consistently throughout participation in the trial. Essential changes are permitted
* If taking PD medications or any nutraceuticals, must be on a stable dose for at least 30 days prior to Screening Visit. Essential changes will be permitted.
* If subject is taking chronic antidepressant or an anxiolytic, must be on a stable dose for at least 90 days prior to Screening. Essential changes will be permitted.

Key Exclusion Criteria:

* Clinical diagnosis of Type 1 or Type 2 Diabetes Mellitus
* Glycated hemoglobin (HbA1c) level ≥ 6.5%
* History of hypoglycemia and/or documented plasma glucose levels of ≤ 50 mg/dL with or without symptoms of hypoglycemia
* Mini-Mental State Exam (MMSE) score of ≤ 24 at Screening
* Positive COVID-19 test at Screening and/or within 30 days of Screening
* Change in or escalation of dose of a chronic therapeutic agent that has the potential to impair cognitive functioning
* Chronic inflammation of nasal cavity that may prevent absorption of study treatments
* Insufficiently controlled respiratory disease (i.e., asthma, COPD).
* History of any significant neurologic or psychiatric disease other than PD
* Current diagnosis of epilepsy and had a history of seizures as an adult within 1 year of Screening, or unexplained recent loss of consciousness, or history of significant head trauma with loss of consciousness
* History of non-lacunar ischemic and/or hemorrhagic stroke
* Unstable or uncontrolled cardiac disease that could expose the subject to additional safety risks
* Use of the following medications: Insulin or any other anti-hyperglycemic agent(s) except if used during isolated gestational diabetes, Supplementation with GSH or any medication shown to increase glutathione, and Beta Blockers

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Verbal Fluency | 24 Weeks
  F, A and S (FAS) words test

SECONDARY OUTCOMES:
Verbal Fluency | 28 Weeks
  Change in verbal fluency as assessed by the FAS test
Motor Function | 24 Weeks
  Change in Timed Up and Go (TUG) test
Motor Function | 24 Weeks
  Change in the updated Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III total score
Motor Function | 24 Weeks
  Change in the updated MDS-UPDRS total score
Motor Function | Week 24
  Change in the Clinical Global Impression (CGI) score
Motor Function | Week 24
  Change in Clinical Impression of Severity Index for Parkinson's Disease (CISI-PD)
Cognitive Function | Week 24
  Change in each of the individual twelve (12) task standardized scores assessed using the Cambridge Brain Sciences (CBS) computerized neuropsychological battery
Non-Motor Function | Week 24
  Change in Hamilton Rating Scale for Depression total score
Patient Reported Outcome | Week 24
  Change in Parkinson's Disease Quality of Life Questionnaire (PDQ-39) assessment
Patient Reported Outcome | Week 24
  Change in the Patient Global Impression (PGI) score

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Institute for Neuroimmune Medicine, Davie, Florida
  - Las Mercedes Medical Research, Hialeah, Florida